CLINICAL TRIAL: NCT00375336
Title: Risk Markers of Coronary Artery Disease Associated With Calcific Aortic Valve Disease
Brief Title: Risk Factors Associated With Calcification of the Aortic Valve
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Ivana Ratajova, Charles University, School of Medicine Plzen
Other Study IDs: IGA MH NR/8306-5
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2008-12

CONDITIONS: Aortic Stenosis; Aortic Sclerosis
Keywords: Aortic valve; Calcification; Endothelial dysfunction; Calcium metabolism; Coronary artery disease
MeSH Terms: conditions — Aortic Valve Stenosis; Calcinosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma specimens retained at -80 deg. C
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients with aortic stenosis (mean transvalvular aortic gradient ≥30 mm Hg) plus angiographically significant coronary artery disease (more than 50% diameter stenosis)
- 2: Patients with nonobstructive aortic sclerosis (mean gradient ≤10 mmHg) plus angiographically significant coronary artery disease (more than 50% diameter stenosis)
- 3: Patients with normal aortic valve plus angiographically significant coronary artery disease (more than 50% diameter stenosis)

SUMMARY:
The purpose of this study is

* to determine the degree of endothelial dysfunction and inflammation in calcific aortic valve disease associated with coronary artery disease(CAD).
* to determine whether there is relationship between calcium metabolism and calcific aortic valve disease associated with CAD.

DETAILED DESCRIPTION:
Cardiovascular disease, mainly coronary artery disease, causes more than one half of deaths in the developed countries. Only recently, calcific aortic valve disease, was proved to belong to the family of atherosclerosis. It is associated with higher cardiovascular morbidity and mortality, the cause of which is not entirely clear. The link to significant coronary artery disease, probably, is of highest importance.

We compare groups of patients with coronary artery disease and calcific stenotic, sclerotic or intact aortic valve. The aim is to assess and compare their risk profile to verify our hypothesis that, within significant coronary artery disease, calcific aortic valve identifies a subgroup of patients with higher cardiovascular risk, assessed by endothelial dysfunction and the two year follow-up of cardiovascular events on optimally set treatment.

Further, we study the possible association of valvular calcification and calcium metabolism in patients with normal kidney function.

ELIGIBILITY:
Inclusion criteria:

* significant stenosis (more than 50% diameter stenosis) of one or more coronary arteries
* aortic sclerosis (group 1) or stenosis (AVA < 1cm2/m2, or mean gradient ≥ 30 mmHg) (group 2) or normal aortic valve (group 3)

Exclusion criteria:

* Rheumatic heart disease (defined as aortic stenosis with commissural fusion + rheumatic mitral valve disease)
* Status post aortic valve replacement
* Congenital complex heart disease (except bicuspid aortic valve)
* Moderate to severe aortic insufficiency (grade > 2/4)
* Marfan syndrome
* Infective endocarditis
* Hypertrophic obstruction cardiomyopathy
* Acute coronary syndrome within less than three months
* Severe heart failure, NYHA class IV
* Severe locomotion disability
* Renal failure requiring dialysis
* Significant systemic disease or other disease severely limiting the patient prognosis (e.g. known cancer, liver cirrhosis)
* Primary hyperparathyroidism
* Patient non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to hospital for evaluation due to common causes like dyspnea, chest pain, fatigue or syncope, who fulfilled the two inclusion criteria: 1/ angiographically significant CAD, and 2/ AS (mean transvalvular aortic gradient ≥30 mm Hg) or nonobstructive aortic sclerosis (mean gradient ≤10 mmHg) or had normal aortic valve as diagnosed by echocardiography.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-01; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Linhartova, MD, PhD, Principal Investigator — Charles University of Prague, School of Medicine Pilsen, Czech Republic; Roman Cerbak, Prof,MD,PhD, Study Chair — Center for Cardiovascular and Transplantation Surgery, Brno, Czech Republic
Locations (1):
- Charles University of Prague, School of Medicine, Plzen, Pilsen, Czechia

REFERENCES:
- [Background] Linhartova K, Filipovsky J, Cerbak R, Sterbakova G, Hanisova I, Beranek V. Severe aortic stenosis and its association with hypertension: analysis of clinical and echocardiographic parameters. Blood Press. 2007;16(2):122-8. doi: 10.1080/08037050701343241. PMID 17612911
- [Background] Ferda J, Linhartova K, Kreuzberg B. Comparison of the aortic valve calcium content in the bicuspid and tricuspid stenotic aortic valve using non-enhanced 64-detector-row-computed tomography with prospective ECG-triggering. Eur J Radiol. 2008 Dec;68(3):471-5. doi: 10.1016/j.ejrad.2007.09.011. Epub 2007 Oct 24. PMID 17961946
- [Background] Linhartova K, Beranek V, Sefrna F, Hanisova I, Sterbakova G, Peskova M. Aortic stenosis severity is not a risk factor for poststenotic dilatation of the ascending aorta. Circ J. 2007 Jan;71(1):84-8. doi: 10.1253/circj.71.84. PMID 17186983
- [Result] Linhartova K, Veselka J, Sterbakova G, Racek J, Topolcan O, Cerbak R. Parathyroid hormone and vitamin D levels are independently associated with calcific aortic stenosis. Circ J. 2008 Feb;72(2):245-50. doi: 10.1253/circj.72.245. PMID 18219161